CLINICAL TRIAL: NCT01289717
Title: Discovery and Validation of Proteogenomic Biomarker Panels in a Prospective Serial Blood & Urine Monitoring Study of Kidney Transplant Recipients - Transplant Proteogenomics
Brief Title: Proteogenomic Biomarker Panels in a Serial Blood & Urine Monitoring Study of Kidney Transplant Recipients
Acronym: PROGENI-KI
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOT-08
Record Dates: First submitted 2011-02-02; First posted 2011-02-04 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Kidney Transplant; Kidney Transplantation
Keywords: biomarkers; proteogenomic profiling; acute rejection; chronic allograft nephropathy/interstitial fibrosis and tubular atrophy
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of blood, urine, and tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is a need to develop blood and/or urine tests that will help to detect early signs of rejection in people who have had kidney transplant. Researchers will examine blood, urine, and tissue samples and try to identify genetic markers for certain conditions like rejection, response to therapy, and scarring of the kidney. By studying gene patterns, researchers hope to be able to diagnose these conditions earlier and improve kidney survival.

DETAILED DESCRIPTION:
Kidney transplantation is a good treatment option for people with kidney disease. However, there is still much to learn about how to best care for the transplanted kidney and keep it working for a long time. One field of interest is how one's cellular make-up might affect the body's immune response (body's natural defense system to illness and foreign things) to a kidney transplant. Cellular tests, like gene expression, help doctors to study a person's cellular traits. Gene expression is when information found in one's DNA is translated into RNA and eventually proteins. These components are present in each of the body's cells. In this study, researchers are trying to learn if certain changes in the RNA and proteins found in blood, urine, or transplant biopsy tissue can detect rejection before injury can occur or become too severe. The blood and urine tests will look for patterns in one's DNA (called genetic markers).

This study will follow subjects for 2 years after transplant. There will be a total of 12 study visits with additional study visits if rejection occurs. The study requires additional samples of blood, urine, and tissue to be collected during routine clinical visits and biopsies (a procedure to remove and examine a small piece of kidney tissue).

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing primary or subsequent deceased-donor or living donor kidney transplantation
* Subject and/or parent guardian must be able to understand and provide informed consent
* Female subjects of childbearing potential must have a negative pregnancy test within 6 weeks of study entry.

Exclusion Criteria:

* Need for combined organ transplantation with an extra-renal organ and/or islet
* Recipient of previous non-renal solid organ and/or islet cell transplantation
* Infection with hepatitis C virus (HCV) or human immunodeficiency virus (HIV)
* Inability or unwillingness of a participant to give written informed consent or comply with study protocol
* Any condition that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing kidney transplantation.
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2011-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Biopsy Proven Acute Rejection (AR)-Clinical and Sub-Clinical), Chronic Allograft Nephropathy/Interstitial Fibrosis and Tubular Atrophy (CAN/IFTA), and Normal Renal Biopsy with Stable, Good Kidney Function | 12 and 24 months

SECONDARY OUTCOMES:
Incidence of Death | Baseline to month 24
Incidence of Graft Loss | Baseline to month 24
Incidence of Opportunistic infections | Baseline to month 24
Incidence of BKV, CMV, and EBV Infection | Baseline to month 24
Incidence of Treated Urinary Tract Infection | Baseline to month 24
Incidence of Malignancy | Baseline to month 24
Changes that Occur in Blood, Urine, and Kidney Tissue Gene Expression Signature | Month 1 to month 24
Changes in Plasma Protein Expression Profile | Month 1 to month 24
Changes in Urine Protein Expression Profile | Month 1 to month 24
Changes in Blood MicroRNA Expression Profile | Month 1 to month 24
Evolution of Gene and Protein Expression Profiles During Response to Therapy for AR | Month 1 to month 24
Evolution of Gene and Protein Expression Profiles During Progression or Regression of CAN/IFTA on Protocol Biopsies | Month 1 to month 24

CONTACTS AND LOCATIONS:
Overall Officials: Michael Abecassis, MD, MBA, Principal Investigator — Northwestern University; John J Friedewald, MD, Study Chair — Northwestern University
Locations (5):
- United States (5):
  - Mayo Clinic, Division of Nephrology, Phoenix, Arizona
  - The Scripps Research Institute, Scripps Center for Organ and Cell Transplantation,, La Jolla, California
  - Northwestern University, Feinberg School of Medicine, Division of Organ Transplantation, Chicago, Illinois
  - The Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Division of Transplant, Charleston, South Carolina

REFERENCES:
- [Background] Kurian SM, Heilman R, Mondala TS, Nakorchevsky A, Hewel JA, Campbell D, Robison EH, Wang L, Lin W, Gaber L, Solez K, Shidban H, Mendez R, Schaffer RL, Fisher JS, Flechner SM, Head SR, Horvath S, Yates JR, Marsh CL, Salomon DR. Biomarkers for early and late stage chronic allograft nephropathy by proteogenomic profiling of peripheral blood. PLoS One. 2009 Jul 10;4(7):e6212. doi: 10.1371/journal.pone.0006212. PMID 19593431
- [Background] Brouard S, Mansfield E, Braud C, Li L, Giral M, Hsieh SC, Baeten D, Zhang M, Ashton-Chess J, Braudeau C, Hsieh F, Dupont A, Pallier A, Moreau A, Louis S, Ruiz C, Salvatierra O, Soulillou JP, Sarwal M. Identification of a peripheral blood transcriptional biomarker panel associated with operational renal allograft tolerance. Proc Natl Acad Sci U S A. 2007 Sep 25;104(39):15448-53. doi: 10.1073/pnas.0705834104. Epub 2007 Sep 14. PMID 17873064
- [Background] Mas VR, Mas LA, Archer KJ, Yanek K, King AL, Gibney EM, Cotterell A, Fisher RA, Posner M, Maluf DG. Evaluation of gene panel mRNAs in urine samples of kidney transplant recipients as a non-invasive tool of graft function. Mol Med. 2007 May-Jun;13(5-6):315-24. doi: 10.2119/2007-00017.Mas. PMID 17622313
- [Background] Muthukumar T, Dadhania D, Ding R, Snopkowski C, Naqvi R, Lee JB, Hartono C, Li B, Sharma VK, Seshan SV, Kapur S, Hancock WW, Schwartz JE, Suthanthiran M. Messenger RNA for FOXP3 in the urine of renal-allograft recipients. N Engl J Med. 2005 Dec 1;353(22):2342-51. doi: 10.1056/NEJMoa051907. PMID 16319383
- [Background] Veronese F, Rotman S, Smith RN, Pelle TD, Farrell ML, Kawai T, Benedict Cosimi A, Colvin RB. Pathological and clinical correlates of FOXP3+ cells in renal allografts during acute rejection. Am J Transplant. 2007 Apr;7(4):914-22. doi: 10.1111/j.1600-6143.2006.01704.x. Epub 2007 Feb 7. PMID 17286616
- [Result] Kurian SM, Williams AN, Gelbart T, Campbell D, Mondala TS, Head SR, Horvath S, Gaber L, Thompson R, Whisenant T, Lin W, Langfelder P, Robison EH, Schaffer RL, Fisher JS, Friedewald J, Flechner SM, Chan LK, Wiseman AC, Shidban H, Mendez R, Heilman R, Abecassis MM, Marsh CL, Salomon DR. Molecular classifiers for acute kidney transplant rejection in peripheral blood by whole genome gene expression profiling. Am J Transplant. 2014 May;14(5):1164-72. doi: 10.1111/ajt.12671. Epub 2014 Apr 11. PMID 24725967
- See also: National Institutes of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Clinical Trials in Organ Transplantation (CTOT) — https://www.ctotstudies.org/